CLINICAL TRIAL: NCT01045395
Title: Efficacy of Two Algae Formulations on Lipid Metabolism, Inflammation and Oxidative Stress Status in Individuals With Psoriasis
Acronym: PCA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Dr. Peter Jones Director Richardson Centre for Functional Foods and Nutraceuticals, Richardson Centre for Functional Foods and Nutraceuticals, University of Manitoba
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: B2008:139
Record Dates: First submitted 2010-01-07; First posted 2010-01-11 (Estimated); Last update posted 2011-03-16 (Estimated); Status verified 2010-01

CONDITIONS: Psoriasis
Keywords: Algae; Psoriasis; Lipid metabolism; Inflammation; Oxidative stress
MeSH Terms: conditions — Psoriasis; Inflammation | interventions — Starch

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Corn starch, 90mg/d (Placebo Comparator): Corn starch, 90mg/d
  Interventions: Dietary Supplement: Corn starch
- Unique Marine Algae Concentrate (UMAC). 90mg/d (Experimental)
  Interventions: Dietary Supplement: Unique Marine Algae Concentrate (UMAC)
- Golden brown algae, 90mg/d (Experimental)
  Interventions: Dietary Supplement: Golden brown algae

INTERVENTIONS:
Dietary Supplement: Corn starch — 90mg/d
  Arms: Corn starch, 90mg/d
Dietary Supplement: Unique Marine Algae Concentrate (UMAC) — 90mg/d
  Arms: Unique Marine Algae Concentrate (UMAC). 90mg/d
Dietary Supplement: Golden brown algae — 90mg/d
  Arms: Golden brown algae, 90mg/d

SUMMARY:
Our overall goal is to evaluate the safety and efficacy of consumption of two algae formulations compared to a placebo on: degree of severity of skin lesions, plasma lipid levels, as well as other health-related markers, in individuals with clinically diagnosed psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Males and females with clinically diagnosed psoriasis
* Plasma LDL-C 80-190 mg/dL, and TG levels below 400 mg/dL.
* Body mass index (BMI) range will be 22 to 32 kg/m2.
* Subjects must demonstrate an ability to understand dietary procedures and be judged as compliant and motivated by the investigators.
* Subjects will be permitted to take stable doses of medications (including drugs for thyroid disease and hypertension)will be permitted if the dose level is maintained stable throughout the study.
* potential subjects must have stable psoriasis and their treatments must remain constant throughout the study.

Exclusion Criteria:

* recent (i.e. less than 3 mo) or chronic use of oral hypolipidemic therapy, including fish oils, or probucol within the last 6 mo
* history of chronic use of alcohol (>2 drinks/d), systemic antibodies, corticosteroids, androgens, or phenytoin
* subjects on anticoagulant therapy (such as warfarin), taking medications and/or natural health products known to affect lipid metabolism (cholestyramine, colestipol, niacin, clofibrate, gemfibrozil, probucol, HMG CoA reductase inhibitors, high dose dietary supplements or fish oil capsules (>4g/day), guggul, lecithin, evening primrose oil within the last six month period will be excluded. In addition, subjects will not be allowed to consume any of these medications during the study
* myocardial infarction, coronary artery bypass, or other major surgical procedures within the last six months
* recent onset and any history of angina, congestive heart failure, heart disease, inflammatory bowel disease, pancreatitis, diabetes, lactose intolerance gastrointestinal, renal, pulmonary, hepatic or biliary disease, or cancer
* moderate or high risk for CAD
* uncontrolled hypertension defined as untreated systolic blood pressure > 160 mmHg and/or diastolic blood pressure > 100 mmHg
* pregnant, breastfeeding, or planning to become pregnant during the course of the trial
* bleeding disorder, anemia, or significant recent blood loss/donation
* allergy/sensitivity to any of the ingredients in the study product or placebo
* chronic user of algal products, fiber laxative (greater than 2 doses/wk), or stimulant laxatives or has a history of eating disorders, exercise greater than 15 miles/wk or 4,000 kcal/wk.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-06 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
A photographic documentation will be carried out quantifying lesion size over at least two body sites. A subjective questionnaire will also be provided to volunteers to enable self-reported evaluation of the extent and degree of discomfort of lesions. | at the beginning and end of each of the three intervention periods
Total cholesterol, LDL- cholesterol, HDL-cholesterol and Triglycerides in plasma, will be determined. | at the beginning and the end of each phase

SECONDARY OUTCOMES:
Vascular cell adhesion molecule-1 (VCAM-1), E-selectin, interleukin-6 (IL-6), IL-10, soluble tumour necrosis factor receptor 2 (sTNFR-2) and soluble cell adhesion molecules (sICAM-1 and sVCAM-1) will be assessed. Lipid peroxidation will also be measured. | at the beginning and the end of each phase

CONTACTS AND LOCATIONS:
Locations (1):
- Ricahrson Centre for Functionl Foods and Nutraceuticals, U of M, Winnipeg, Manitoba, Canada